CLINICAL TRIAL: NCT05575999
Title: Pain Management in Cardiac Implantable Electronic Device Insertion; Effectiveness of Bupivacaine, Ketorolac, Ketamine, vs Bupivacaine Alone in Reducing Postoperative Pocket Pain
Brief Title: Effectiveness of Bupivacaine, Ketorolac, Ketamine, vs Bupivacaine Alone in Reducing Postoperative Pocket Pain
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Cardiac Arrhythmia Service, Loma Linda University Health, Loma Linda, CA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCHRRF-PAINFREE POCKET-0016
Record Dates: First submitted 2022-09-16; First posted 2022-10-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-10

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine Alone (Other): This is the control group of patients receiving 20 cc of 0.5% bupivacaine (Bupivacaine HCL 100 mg [5mg/ml] alone. The dose and number of doses of the medicines will be adjusted as per discretion of the operator.
  Interventions: Drug: Bupivacaine alone OR Bupivacaine-Ketorolac-Ketamine (BKK) Combination
- Bupivacaine-Ketorolac-Ketamine (BKK) Combination (Experimental): This is the intervention group of patients receiving 20 cc combination of BKK (Bupivacaine HCl 60 mg [3 mg/mL], Ketorolac Tromethamine 24 mg [1.2mg/mL], Ketamine HCl 24 mg [1.2 mg/mL]).The dose and number of doses of the medicines will be adjusted as per discretion of the operator.
  Interventions: Drug: Bupivacaine alone OR Bupivacaine-Ketorolac-Ketamine (BKK) Combination

INTERVENTIONS:
Drug: Bupivacaine alone OR Bupivacaine-Ketorolac-Ketamine (BKK) Combination — The plan will be to stratify patients in two groups: intervention group receiving 20 cc combination of BKK (Bupivacaine HCl 60 mg [3 mg/mL], Ketorolac Tromethamine 24 mg [1.2mg/mL], Ketamine HCl 24 mg [1.2 mg/mL]) vs the control group receiving 20 cc of 0.5% bupivacaine (Bupivacaine HCL 100 mg [5mg/ml]. The dose can be repeated multiple times during the procedure as per operator's discretion. The patients will be further stratified into sub-groups based on type of procedure they had undergone. Analgesia/anesthesia strategy will be local infiltration of the drug along with a sedating agent based on institutional standard of care. The dose of the medicines will be adjusted as per discretion of the operator to maintain adequate anesthesia/analgesia during and after the procedure.

SUMMARY:
Bupivacaine is the most widely used local anesthetic agent across majority of the Cardiac Implantable Electronic device (CIED) implant procedures in the United States. It is hypothesized that the combination of Bupivacaine-Ketorolac-Ketamine (BKK) is more effective in alleviating perioperative and postoperative pain as compared to the use of bupivacaine alone.

A few studies have been done to look for the effectiveness of BKK in abdominal surgical procedures. However, no study has been done to evaluate its efficacy and effectiveness in patients undergoing CIED insertion.

DETAILED DESCRIPTION:
Bupivacaine is a widely used local anesthetic and is often administered by spinal injection prior to major surgical procedures. Ketorolac is a potent NSAID which is used for the short-term relief of moderate to severe pain. It's used for long term duration is generally limited due to its potential to cause GI ulcers/perforation and renal failure. A single dose of perioperative Ketorolac has been found to be effective in reducing opioid consumption. Ketamine is NMDA receptor antagonist and is used for its anesthetic, analgesic, and psychotomimetic effects. It is primarily used for induction and maintenance of anesthesia and induces a trance like state providing pain relief, sedation, and amnesia.

Although an effective local anesthetic agent, bupivacaine has weak analgesic effect and is used in combination with several analgesic agents for effective perioperative and postoperative analgesia. A common drug used in this analgesic regimen usually includes opioids such as morphine, oxycodone, and fentanyl. Over the last few decades the United States has witnessed an opioid epidemic and post-surgical opioid prescription is one of the major contributors of this epidemic. An opioid free combination of Bupivacaine-Ketorolac-Ketamine (BKK) is thought to be effective in alleviating perioperative and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients
* Patients older than 18 years of age
* Patients undergoing new CIED (ICD, pacemaker, CRT-D or CRT-P)
* Patients willing to participate in the study

Exclusion Criteria:

* Patients with prior history of allergic reaction to any component of the drug; bupivacaine, ketorolac, or ketamine
* Pregnant or breastfeeding patients
* Prisoners
* Patients younger than 18 years of age
* Patients not willing to participate in the study
* Patients deemed not suitable or unstable for the study as per physician's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparative efficacy/superiority of BKK compared to bupivacaine alone in reducing the pain intensity | Upto 1 week
  The goal of this prospective open label study is to demonstrate a comparative efficacy/superiority of BKK compared to bupivacaine alone in reducing the pain intensity. Patient's pain will be assessed using a Visual Analog Scale either through a telephone call from the research team or via clinic follow-up visit. The visual analog scale (VAS) determines pain from 0 to 10 with 0 indicating no pain (Better outcome) and 10 indicating worse pain in their life indicating (worse outcome).
Comparative efficacy/superiority of BKK compared to bupivacaine alone in providing comfort | Upto 1 week
  The goal of this prospective open label study is to demonstrate a comparative efficacy/superiority of BKK compared to bupivacaine alone in providing comfort. Patient's comfort will be assessed using a verbal rating score either through a telephone call from the research team or via clinic follow-up visit. The comfort score determines patients comfort from 0 to 100 with 0 indicating extremely uncomfortable (Worse outcome) and 100 indicating extremely comfortable (Better outcome).
Comparative efficacy/superiority of BKK compared to bupivacaine alone in Quality of Life (QoL) | Upto 1 week
  The goal of this prospective open label study is to demonstrate a comparative efficacy/superiority of BKK compared to bupivacaine alone in Quality of Life. Patient's Quality of Life will be assessed using a QoL score (EQ5-5D-5L) either through a telephone call from the research team or via clinic follow-up visit. The Quality of life questionnaire (EQ-5D-5L) has five response levels : no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5), with low values suggesting better outcomes and higher values suggesting worse outcomes.

SECONDARY OUTCOMES:
Hospital readmission rates | Until 7 days (Until the end of the sutdy)
  Hospital readmission rates due to device implantation related pain or surgical site infection will be analyzed.
Adverse Effects | Until 7 days (Until the end of the sutdy)
  Rates of adverse effects, including allergic reaction, worsening of the renal function, presyncope/syncope, HTN, drug-drug interaction or any patient reported side effects will be analyzed.
Cost comparison of medications | Upto 1 week
  Cost of medications will be compared.
Amount of pain medication used | Upto 1 week
  Amount of pain medication used will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (3):
- United States (3):
  - Loma Linda University Health, Loma Linda, California
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mariano ER, Dickerson DM, Szokol JW, Harned M, Mueller JT, Philip BK, Baratta JL, Gulur P, Robles J, Schroeder KM, Wyatt KEK, Schwalb JM, Schwenk ES, Wardhan R, Kim TS, Higdon KK, Krishnan DG, Shilling AM, Schwartz G, Wiechmann L, Doan LV, Elkassabany NM, Yang SC, Muse IO, Eloy JD, Mehta V, Shah S, Johnson RL, Englesbe MJ, Kallen A, Mukkamala SB, Walton A, Buvanendran A. A multisociety organizational consensus process to define guiding principles for acute perioperative pain management. Reg Anesth Pain Med. 2022 Feb;47(2):118-127. doi: 10.1136/rapm-2021-103083. Epub 2021 Sep 22. PMID 34552003
- [Background] De Oliveira GS Jr, Agarwal D, Benzon HT. Perioperative single dose ketorolac to prevent postoperative pain: a meta-analysis of randomized trials. Anesth Analg. 2012 Feb;114(2):424-33. doi: 10.1213/ANE.0b013e3182334d68. Epub 2011 Sep 29. PMID 21965355
- [Background] Wolfe RC, Spillars A. Local Anesthetic Systemic Toxicity: Reviewing Updates From the American Society of Regional Anesthesia and Pain Medicine Practice Advisory. J Perianesth Nurs. 2018 Dec;33(6):1000-1005. doi: 10.1016/j.jopan.2018.09.005. No abstract available. PMID 30449428
- [Background] Nair GM, Birnie DH, Sumner GL, Krahn AD, Healey JS, Nery PB, Kalfon E, Verma A, Ayala-Paredes F, Coutu B, Becker G, Philippon F, Eikelboom J, Sandhu RK, Sapp J, Leather R, Yung D, Thibault B, Simpson CS, Ahmad K, Sturmer M, Kavanagh K, Crystal E, Wells GA, Essebag V; BRUISE CONTROL Investigators. Post-operative pain following cardiac implantable electronic device implantation: insights from the BRUISE CONTROL trials. Europace. 2021 May 21;23(5):748-756. doi: 10.1093/europace/euaa349. PMID 33367623
- [Background] Neuman MD, Bateman BT, Wunsch H. Inappropriate opioid prescription after surgery. Lancet. 2019 Apr 13;393(10180):1547-1557. doi: 10.1016/S0140-6736(19)30428-3. PMID 30983590
- [Background] Clerc S, Vuilleumier H, Frascarolo P, Spahn DR, Gardaz JP. Is the effect of inguinal field block with 0.5% bupivacaine on postoperative pain after hernia repair enhanced by addition of ketorolac or S(+) ketamine? Clin J Pain. 2005 Jan-Feb;21(1):101-5. doi: 10.1097/00002508-200501000-00012. PMID 15599137